CLINICAL TRIAL: NCT04540627
Title: A Double-Blind, Randomised, Placebo-Controlled Exploratory Study to Estimate the Prophylactic Efficacy of Palivizumab in Healthy Adult Participants Inoculated With Respiratory Syncytial Virus (RSV)
Brief Title: Exploratory Study to Estimate the Prophylactic Efficacy of Palivizumab in Healthy Adult Participants Inoculated With RSV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MB05-P-01-20
Record Dates: First submitted 2020-07-24; First posted 2020-09-07 (Actual); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Healthy Adult Participants
MeSH Terms: interventions — Palivizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Sodium Chloride 0.9% Solution (Normal Saline)
  Interventions: Drug: Placebo; Other: RSV-A Memphis 37b virus
- Palivizumab (Synagis™) (Active Comparator): Sterile vial 50mg/0.5mL
  Interventions: Drug: Palivizumab; Other: RSV-A Memphis 37b virus

INTERVENTIONS:
Drug: Palivizumab — Liquid solution in sterile water for injection (final concentration of 20mg/mL), intravenous infusion, single dose of 8mg/kg or 15mg/kg, administered at a rate of 1mL/min
  Other Names: Synagis™
  Arms: Palivizumab (Synagis™)
Drug: Placebo — Sodium Chloride 0.9% Solution (Normal Saline), intravenous infusion, single dose of 0mg/Kg, administered at a rate of 1mL/min
  Arms: Placebo
Other: RSV-A Memphis 37b virus — Single Intranasal Virus Dose (challenge dose is approximately 4.5log10 PFU)

SUMMARY:
Double-Blind, Randomised, Placebo-Controlled Exploratory Study to Estimate the Prophylactic Efficacy of Palivizumab in Healthy Adult Participants Inoculated with Respiratory Syncytial Virus (RSV).

DETAILED DESCRIPTION:
As no data exists for Palivizumab in the RSV human challenge model, this exploratory study is therefore planned to establish the margins of effect and variance of prophylactically administered Palivizumab within the RSV-A Memphis 37b challenge model in healthy adult volunteers.

The study will be performed in adults aged 18-55 years, in two parts.

• Part 1: All participants will be administered Palivizumab (8mg/Kg, intravenously). Pharmacokinetic (PK), safety will be measured.

If there are no safety concerns in Part 1, and PK analysis of Palivizumab treated participants confirm the modelling of 8mg/Kg to be appropriate, Part 2 will commence with the planned 8mg/Kg treatment dose. However, if PK analysis of Part 1 suggests that 8mg/kg may be insufficient dose to provide suitable efficacious coverage in Part 2, then Part 2 will proceed with a dose of 15mg/Kg.

• Part 2: Participants will be either administered Palivizumab (8mg/Kg or 15mg/Kg, as determined in Part ) or a placebo and they will subsequently be challenged with an RSV-A strain (Memphis 37b). The margin of effect and variance between groups will be measured, as well as safety and reactogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent document signed and dated by the participant and the Investigator.
2. Aged between 18 and 55 years old on the day of signing the consent form.
3. In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that will interfere with participant safety, as defined by medical history, physical examination, (including vital signs), Electrocardiogram (ECG), and routine laboratory tests as determined by the Investigator.
4. A documented medical history prior to enrolment.
5. The following criteria are applicable to female participants participating in the study.

   1. Females of childbearing potential must have a negative pregnancy test prior to enrolment.
   2. Females of non-childbearing potential:

   <!-- -->

   1. Post- menopausal females; defined as having a history of amenorrhea for >12 months with no alternative medical cause, and /or by Follicle stimulating hormone (FSH) level >40mIU/mL, confirmed by laboratory
   2. Documented status as being surgically sterile (e.g. tubal ligation, hysterectomy, bilateral salpingectomy and bilateral oophorectomy).
6. The following criteria apply to female and male participants:

   1. Female participants of childbearing potential must use one form of highly effective contraception. Hormonal methods must be in place from at least 2 weeks prior to the first study visit. The contraception use must continue until 30 days after the date of viral challenge/last dosing with IMP (whichever occurs last). Highly effective contraception is as described below:

   <!-- -->

   1. Established use of hormonal methods of contraception described below (for a minimum of 2 weeks prior to the first study visit). When hormonal methods of contraception are used, male partners are required to use a condom with a spermicide:

1. Oral 2. Intravaginal 3. Transdermal b. Intrauterine device (IUD) c. Intrauterine hormone-releasing system (IUS) d. Bilateral tubal ligation e. Male sterilisation (with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate) where the vasectomised male is the sole partner for that woman.

f. True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.

b) Male participants must agree to the contraceptive requirements below at entry to quarantine and continuing until 90 days after the date of Viral challenge / last dosing with the investigational medicinal product (IMP) (whichever occurs last):

1. Use a condom with a spermicide to prevent pregnancy in a female partner or to prevent exposure of any partner (male and female) to the IMP.
2. Male sterilisation with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate (please note that the use of condom with spermicide will still be required to prevent partner exposure). This applies only to males participating in the study
3. In addition, for female partners of childbearing potential, that partner must use another form of contraception such as one of the highly effective methods mentioned above for female participants.
4. True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.

c) In addition to the contraceptive requirements above, male participants must agree not to donate sperm following discharge from quarantine until 90 days after the date of Viral Challenge/last dosing with IMP (whichever occurs last).

7. For Part 2 of the study: Sero-suitable to the challenge virus, as defined in the study Analytical Plan.

Exclusion Criteria:

Medical History

1. History of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract infection within 4 weeks prior to the first study visit.
2. a) Any history or evidence of any other clinically significant or currently active systemic comorbidities including psychiatric disorders (includes participants with a history of depression and/or anxiety).

   b) And/or other major disease that, in the opinion of the Investigator, may put the participant at undue risk, or interfere with a participant completing the study and necessary investigations.

   The following conditions apply:

   • Participants with clinically mild atopic eczema/atopic dermatitis and clinically mild psoriasis may be included at the Investigator's discretion (e.g., if small amounts of regular topical steroids are used, no eczema in cubital fossa; moderate to large amounts of daily dermal corticosteroids is an exclusion).
   * Rhinitis (including hay fever) which is clinically active or history of moderate to severe rhinitis, or history of seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on an at least weekly basis, within 30 days of admission to quarantine will be excluded. Participants with a history of currently inactive rhinitis (within the last 30 days) or mild rhinitis may be included at the PI's discretion.
   * Participants with a physician diagnosed underactive thyroid who have been controlled on treatment for at least 6 months with evidence of a normal thyroid function test (TFT) can be included at the discretion of the PI.
   * Any concurrent serious illness including history of malignancy that may interfere with the aims of the study or a participant completing the study. Basal cell carcinoma within 5 years of initial diagnosis or with evidence of recurrence is also an exclusion.

     o Participants with a history of psychiatric illness including depression and/or anxiety of any severity within the last 2 years can be included if the Patient Health Questionnaire (PHQ-9) and / or the Generalised Anxiety Disorder Questionnaire (GAD-7) is less than or equal to 4. Participants with a PHQ-9 or GAD-7 score of between 5 and 9 may be included following consultation with a Senior Physician (Clinical Lead for Screening) who may advise further consultation with the PI.

     o Participants reporting physician diagnosed migraine can be included provided there are no associated neurological symptoms such as hemiplegia or visual loss. Cluster headache/migraine or prophylactic treatment for migraine is an exclusion.
     * Participants with physician diagnosed mild Irritable Bowel Syndrome (IBS) not requiring regular treatment can be included at the discretion of the PI.
3. Participants who have smoked ≥ 10 pack years at any time [10 pack years is equivalent to one pack of 20 cigarettes a day for 10 years]).
4. A total body weight ≤ 50 kg and Body Mass Index (BMI) ≤18 kg/m2 and ≥30kg/m2
5. Females who:

   1. Are breastfeeding, or
   2. Have been pregnant within 6 months prior to the study.
6. History of anaphylaxis-and/or a history of severe allergic reaction or significant intolerance to any food or drug, as assessed by the PI.
7. Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
8. a) For Part 2 of the study: Any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx that may interfere with the aims of the study and in particular any of the nasal assessments or viral challenge, (historical nasal polyps can be included, but large nasal polyps causing current and significant symptoms and/or requiring regular treatments in the last month will be excluded).

   b) Any clinically significant history of epistaxis (large nosebleeds) within the last 3 months of the first study visit and/or history of being hospitalized due to epistaxis on any previous occasion.

   c) Any nasal or sinus surgery within 3 months of the first study visit. Prior or Concomitant Medications and Assessments
9. For Part 2 of the study:

   1. Evidence of vaccinations within the 4 weeks prior to the planned date of viral challenge/first dosing with IMP (whichever occurs first).
   2. Intention to receive any vaccination(s) before the last day of Follow-up. (NB. No travel restrictions will apply after the Day 28 (±3 days) Follow-up Visit).
10. Receipt of blood or blood products, or loss (including blood donations) of 470 mL or more of blood during the 3 months prior to the planned date of viral challenge/first dosing with IMP (whichever occurs first) or planned during the 3 months after the final visit.
11. a) Receipt of any investigational drug within 3 months prior to the planned date of viral challenge/first dosing with IMP (whichever occurs first).

    b) Receipt of three or more investigational drugs within the previous 12 months prior to the planned date of viral challenge/first dosing with IMP (whichever occurs first).

    For Part 2 of the study:

    c) Prior inoculation with a virus from the same virus-family as the challenge virus.

    d) Prior participation in another human viral challenge study with a respiratory virus in the preceding 3 months, taken from the date of viral challenge in the previous study to the date of expected viral challenge in this study
12. a) Confirmed positive test for drugs of abuse on first study visit. One repeat test allowed at PI discretion.

    b) History or presence of alcohol addiction, or excessive use of alcohol (weekly intake in excess of 28 units alcohol; 1 unit being a half glass of beer, a small glass of wine or a measure of spirits), or excessive consumption of xanthine containing substances (e.g. daily intake in excess of 5 cups of caffeinated drinks e.g. coffee, tea, cola).
13. For Part 2 of the study:

    A forced expiratory volume in 1 second (FEV1) < 80%.
14. Positive human immunodeficiency virus (HIV), active hepatitis A (HAV), B (HBV), or C (HCV) test.

    Other
15. Those employed or immediate relatives of those employed at hVIVO or the Sponsor.
16. Any other finding that, in the opinion of the Investigator, deems the participant unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sungeen Hill, MD, Principal Investigator — hVIVO Services Limited
Locations (1):
- hVIVO Services Limited, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 2 parts: Part 1 (PK sentinel part) and Part 2 (viral challenge part).
  Part 1: Open-label. This part of the study was used to determine the dose of Palivizumab IV for Part 2 (8 or 15 mg/kg).
  Part 2: Double-blind, randomized, and placebo-controlled. Participants received a single IV dose of either Palivizumab (8 mg/kg, as finally determined in Part 1) or a placebo and were subsequently challenged with an RSV-A strain.
Groups:
- Open-label Palivizumab (Part 1): Sterile vial 50mg/0.5mL
  Palivizumab: Liquid solution in sterile water for injection (final concentration of 20mg/mL), intravenous infusion, single dose of 8mg/kg, administered at a rate of 1mL/min
- Double-blind Placebo (Part 2): Sodium Chloride 0.9% Solution (Normal Saline)
  Placebo: Sodium Chloride 0.9% Solution (Normal Saline), intravenous infusion, single dose of 0mg/Kg, administered at a rate of 1mL/min
  RSV-A Memphis 37b virus: Single Intranasal Virus Dose (challenge dose is approximately 4.5log10 PFU)
- Double-blind Palivizumab (Synagis™) (Part 2): Sterile vial 50mg/0.5mL
  Palivizumab: Liquid solution in sterile water for injection (final concentration of 20mg/mL), intravenous infusion, single dose of 8mg/kg, administered at a rate of 1mL/min
  RSV-A Memphis 37b virus: Single Intranasal Virus Dose (challenge dose is approximately 4.5log10 PFU)
Period: Open-label Treatment: PK Sentinel
Arm/Group | Open-label Palivizumab (Part 1) | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Started | 6 (Participants were not enrolled in this arm in the double-blind period.) | 0 (Participants were not enrolled in this arm in the open-label period.) | 0 (Participants were not enrolled in this arm in the open-label period.)
Completed | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Double-blind Treatment: Viral Challenge
Arm/Group | Open-label Palivizumab (Part 1) | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Started | 0 (Participants were not enrolled in this arm in the double-blind period.) | 25 (Participants were not enrolled in this arm in the open-label period.) | 25 (Participants were not enrolled in this arm in the open-label period.)
Completed | 0 | 25 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-label Palivizumab (Part 1) | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2) | Total
Number analyzed (Participants) | 6 | 25 | 25 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.67 (2.58) | 28.16 (6.30) | 26.76 (5.83) | 26.86 (4.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 12 | 5 | 19
  Male | 4 | 13 | 20 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 4 | 23 | 20 | 47
  More than one race | 2 | 2 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Serum Concentrations (Cmax) for Open-label Palivizumab (Part 1) on Day 12.
Description: The PK assessment up to and including Day 12 exposure was used as a decision information for the dose to be given to participants in Part 2. Pharmacokinetic exposure data from at least 5 out of 6 participants were required for dose decision making with a projected exposure of ≥40 μg/mL on Day 12 according to the protocol.
  This was achieved after administration of a single IV dose of Palivizumab at 8 mg/kg. Therefore, a dose of 8 mg/kg was chosen for Part 2.
Time Frame: In Part 1: before the start of infusion; at end of infusion,15 minutes and 0.5, 1, 4, 8, and 12 hours after infusion; and at 1, 2, 3, 7, and 12 days after infusion.
Population: All participants treated had at least 1 post-dose PK result; therefore, all participants were included in the PK analysis population. One participant had an interrupted IV infusion of Palivizumab but received the complete dose of 8 mg/kg.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Open-label Palivizumab (Part 1) | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 6 | 0 | 0
μg/mL | 71.2 (6.11) |  |

2. Primary Outcome: Area Under the Viral Load-time Curve (VL-AUC) as Determined by Polymerase Chain Reaction (qRT-PCR) on Nasal Samples, for Double-blind Palivizumab or Placebo (Part 2).
Description: RSV viral load of RSV-A Memphis 37b as determined by qRT-PCR on nasal samples collected twice daily: Assessment of the Area under the viral load-time curve (VL-AUC)
Time Frame: From two days post viral challenge (Day 2) to the end of quarantine (Day 12) in Part 2 on nasal samples collected twice daily.
Population: The evaluable population includes 49 participants. All participants in this population received study intervention, were inoculated with challenge virus, and completed quarantine. One Palivizumab-treated participant was excluded from the evaluable population because the participant had not completed the quarantine period.
Measure: Mean (Standard Deviation); unit: Log10 copies*day/mL
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Log10 copies*day/mL | 11.68 (15.36) | 9.94 (12.38)
Statistical Analysis 1: Comparison: Double-blind Placebo (Part 2) vs Double-blind Palivizumab (Synagis™) (Part 2); Test type: Superiority; p = 0.5802, Wilcoxon (Mann-Whitney)

3. Primary Outcome: qRT-PCR Peak Viral Load for Double-blind Palivizumab or Placebo (Part 2).
Description: Peak viral load of RSV-A Memphis 37b as determined by qRT-PCR on nasal samples collected twice daily.
Time Frame: From two days post viral challenge (Day 2) to the end of quarantine (Day 12) in Part 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Log10 copies/mL | 3.66 (2.42) | 3.11 (2.65)
Statistical Analysis 1: Comparison: Double-blind Placebo (Part 2) vs Double-blind Palivizumab (Synagis™) (Part 2); Test type: Superiority; p = 0.4868, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Area Under the Viral Load-time Curve (VL-AUC) as Determined by Cell Culture on Nasal Samples, for Double-blind Palivizumab (Part 2).
Description: RSV Viral Load of RSV-A Memphis 37b as Determined by Cell Culture on Nasal Samples collected twice daily: Area under the viral load-time curve (VL-AUC) of RSV-A Memphis 37b
Time Frame: as for outcome 2
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: Log10 PFU*day/mL
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 22 | 22
Log10 PFU*day/mL | 2.05 (5.29) | 1.64 (3.43)
Statistical Analysis 1: Comparison: Double-blind Placebo (Part 2) vs Double-blind Palivizumab (Synagis™) (Part 2); Test type: Superiority; p = 0.2681, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Cell Culture Peak Viral Load for Double-blind Palivizumab or Placebo (Part 2).
Description: Peak Viral Load of RSV-A Memphis 37b as Determined by Cell Culture on Nasal Sample
Time Frame: From Day 2 to Day 12 in Part 2
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: Log10 PFU/mL
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Log10 PFU/mL | 0.60 (1.47) | 0.88 (1.41)
Statistical Analysis 1: Comparison: Double-blind Placebo (Part 2) vs Double-blind Palivizumab (Synagis™) (Part 2); Test type: Superiority; p = 0.2431, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants With Laboratory-confirmed Infection of RSV-A Memphis 37b in Nasal Samples (Variant 1) for Double-blind Palivizumab or Placebo (Part 2).
Description: Percentage of Participants Infected Post-viral Challenge (Infectivity Status and Rate): occurrence of at least 2 positive "quantifiable" qRT-PCR measurements in nasal samples.
  Laboratory-confirmed infection (variant 1): At least 2 positive quantifiable detections by viral load qRT-PCR assay specific for the challenge virus, reported within 4 consecutive scheduled assessments and from 2 independent samples from Day 2 until discharge and/or 1 positive detection by viral load qRT-PCR assay, specific for the challenge virus, in which an aliquot of the same sample has also tested positive in a viral culture assay appropriate for detecting the challenge virus from Day 2 until discharge.
Time Frame: From Day 2 to Day 12 in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Participants | 13 | 12

7. Secondary Outcome: Number of Participants With Laboratory-confirmed Infection of RSV-A Memphis 37b in Nasal Samples (Variant 2), for Double-blind Palivizumab or Placebo (Part 2).
Description: Percentage of Participants Infected Post-viral Challenge (Infectivity Status and Rate): Occurrence of at least 2 positive "detectable" qRT-PCR measurements in nasal samples.
  Laboratory-confirmed infection (variant 2): At least 2 positive detectable assessments by viral load qRT-PCR assay specific for the challenge virus, reported within 4 consecutive scheduled assessments and from 2 independent samples from Day 2 until discharge and/or 1 positive detection by viral load qRT-PCR assay, specific for the challenge virus, in which an aliquot of the same sample has also tested positive in a viral culture assay appropriate for detecting the challenge virus from Day 2 until discharge.
Time Frame: From Day 2 to Day 12 in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Participants | 15 | 15

8. Secondary Outcome: Viral Shedding of RSV-A Memphis 37b in Nasal Samples in Terms of Duration, for Double-blind Palivizumab or Placebo (Part 2).
Description: Estimation of the duration of viral shedding by the number of days with quantifiable qRT-PCR measurements in nasal samples starting 2 days post viral challenge (Day 2) up to the end of quarantine.
Time Frame: From Day 2 to Day 12 in Part 2
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 23
days | 2.84 (3.01) | 2.61 (2.98)

9. Secondary Outcome: Viral Shedding of RSV-A Memphis 37b in Nasal Samples in Terms of Time to Peak Viral Load, for Double-blind Palivizumab or Placebo (Part 2).
Description: Estimation of the duration of viral shedding by the time to peak viral load of RSV by quantifiable qRT-PCR.
Time Frame: From Day 2 to Day 12 in Part 2
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 22 | 16
days | 7.21 (2.98) | 7.03 (2.35)

10. Secondary Outcome: Viral Shedding of RSV-A Memphis 37b in Nasal Samples in Terms of Peak Viral Load, for Double-blind Palivizumab or Placebo (Part 2).
Description: Peak viral load of RSV-A Memphis 37b as defined by the maximum viral load determined by quantifiable qRT PCR measurements in nasal samples starting 2 days post viral challenge (Day 2) up to the end of quarantine.
Time Frame: From Day 2 to Day 12 in Part 2
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Log10 copies/mL | 3.66 (2.42) | 3.11 (2.65)
Statistical Analysis 1: Comparison: Double-blind Placebo (Part 2) vs Double-blind Palivizumab (Synagis™) (Part 2); Test type: Superiority; p = 0.4868, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Total Symptom Score (TSS)-Time Curve (AUC) Collected Daily in the Participant Symptom Diary Card
Description: Mean TSS values (collected daily in the symptom diary card) over time. Symptoms were collected using the hVIVO (services provider) symptom diary card. Several symptoms (such as runny nose, sore throat, earache, etc) in the 13-item questionnaire were graded on a scale of 0-3 (grade 0: No symptoms; grade 1: just noticeable; grade 2: clearly bothersome from time to time but does not interfere with me doing my normal daily activities; grade 3: Quite bothersome most or all of the time, and it stops me participating in activities). Shortness of breath and wheeze have an additional grade 4: Symptoms at rest. The total symptom score (TSS) was determined as the sum of the symptom scores ranging from 0.0 (min) to 41(max) [or a maximum of 41x11.33=464.67 depending on what the reviewer is asking] using a 13-items self-reported diary card. 11.33 is the number of days symptom diary cards were included (Day +1 morning dairy card to Day 12 morning diary card). Higher scores mean worse outcome.
Time Frame: as for outcome 2
Population: Evaluable population
Measure: Mean (Standard Error); unit: Total Symptom Score scale-points*day
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Total Symptom Score scale-points*day | 13.84 (14.72) | 7.27 (9.03)

12. Secondary Outcome: Peak Symptom Scores
Description: Peak symptom scores for symptoms collected daily in the participant symptom diary card.
  Symptoms (such as runny nose, sore throat, earache, etc) were collected using the 13-item hVIVO symptom questionnaire and were graded on a scale of 0-3 (grade 0: No symptoms; grade 1: just noticeable; grade 2: clearly bothersome from time to time but does not interfere with me doing my normal daily activities; grade 3: Quite bothersome most or all of the time, and it stops me participating in activities). Shortness of breath and wheeze have an additional grade 4: Symptoms at rest. The total symptom score (TSS) was determined as the sum of the symptom scores ranging from 0.0 (min) to 41(max) [or a maximum of 41x11.33=464.67 depending on what the reviewer is asking] using a 13-items self-reported diary card. 11.33 is the number of days symptom diary cards were included (Day +1 morning dairy card to Day 12 morning diary card). Higher scores mean worse outcome.
Time Frame: From Day 2 to Day 12 in Part 2
Population: Evaluable population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
score on a scale | 4.16 (3.45) | 2.54 (3.32)
Statistical Analysis 1: Comparison: Double-blind Placebo (Part 2) vs Double-blind Palivizumab (Synagis™) (Part 2); Test type: Superiority; p = 0.0403, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Total Weight of Nasal Discharge Produced
Description: Nasal Discharge Collection from Paper Tissues by means of the total weight of nasal discharge produced.
Time Frame: From Day 1 to Day 12 in Part 2
Population: Evaluable population
Measure: Mean (Standard Error); unit: g
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 23 | 21
g | 22.23 (41.52) | 7.66 (14.92)

14. Secondary Outcome: Total Number of Tissues Used by Participants
Description: Nasal Discharge Collection from Paper Tissues by means of the total number of tissues used.
Time Frame: From Day 1 to Day 12 in Part 2
Population: Evaluable population
Measure: Mean (Standard Error); unit: tissues
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
tissues | 32.04 (42.74) | 20.38 (21.88)

15. Secondary Outcome: Number of Participants With Laboratory-confirmed Virus-like Illness (Variant 1) Using Viral Shedding Variant 1, for Double-blind Palivizumab or Placebo (Part 2).
Description: Illness Post-viral challenge measured by means of the proportion of participants with any symptom ≥grade 1 for the evaluable population.
Time Frame: From Day 2 to Day 12 in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Participants | 11 | 5

16. Secondary Outcome: The Occurrence of Laboratory-confirmed Virus-like Illness (Variant 1) Using Viral Shedding Variant 2, for Double-blind Palivizumab or Placebo (Part 2).
Description: as for outcome 15
Time Frame: From Day 2 to Day 12 in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Participants | 11 | 5

17. Secondary Outcome: The Occurrence of Laboratory-confirmed Virus-like Illness (Variant 2) Using Viral Shedding Variant 1, for Double-blind Palivizumab or Placebo (Part 2).
Description: as for outcome 15
Time Frame: From Day 2 to Day 12 in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Participants | 13 | 11

18. Secondary Outcome: The Occurrence of Laboratory-confirmed Virus-like Illness (Variant 2) Using Viral Shedding Variant 2, for Double-blind Palivizumab or Placebo (Part 2).
Description: as for outcome 15
Time Frame: From Day 2 to Day 12 in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25 | 24
Participants | 15 | 14

19. Secondary Outcome: Cmax
Description: Evaluation of Palivizumab PK levels throughout the study, by means of Cmax after intravenous administration of Palivizumab.
Time Frame: Before the start of infusion; at end of infusion, 15 minutes and 0.5, 1, 4, 8, and 12 hours after infusion; and at 1, 2, 3, 7 and 12 days after infusion (Part 1) or at 1, 2, 3, 7, 13, 21, and 29 days after infusion (Part 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Open-label Palivizumab (Part 1) | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 5 | 0 | 23
μg/mL | 262 (35.6) |  | 283 (46.5)

20. Secondary Outcome: Tmax
Description: Palivizumab PK levels throughout the study, by means of Tmax after intravenous administration of Palivizumab.
Time Frame: Before the start of infusion; at end of infusion, 15 minutes and 0.5, 1, 4, 8, and 12 hours after infusion; and at 1, 2, 3, 7, and 12 days after infusion (Part 1) or at 1, 2, 3, 7, 13, 21, and 29 days after infusion (Part 2)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Groups:
- Open-label Palivizumab (Part 1): Sterile vial 50mg/0.5mL
  Palivizumab: Liquid solution in sterile water for injection (final concentration of 20mg/mL), intravenous infusion, single dose of 8mg/kg or 15mg/kg, administered at a rate of 1mL/min
Arm/Group | Open-label Palivizumab (Part 1) | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 5 | 0 | 23
hours | 0.90 [0.57 to 1.70] |  | 0.92 [0.53 to 1.77]

21. Secondary Outcome: Safety Adults: Number of Participants With Adverse Events (AEs)
Description: Incidence of AEs, treatment-emergent AEs (TEAEs), serious AEs (SAEs) and; drug-related or challenge-virus related TEAEs and SAEs
Time Frame: From Day 1 to Day 18 in Part 1 and from Day 1 to Day 28 in Part 2
Population: Safety analysis population: All participants randomly assigned to study intervention and who took a dose of study intervention, regardless of whether they received the challenge virus or not.
Measure: Number; unit: participants
Arm/Group | Open-label Palivizumab (Part 1) | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 6 | 25 | 25
participants
  Any AE | 0 | 12 | 14
  Any TEAE | 0 | 12 | 14
  Any TEAE related to the study drug | 0 | 1 | 4
  Any TEAE related to the challenge virus | 0 | 5 | 8
  Any SAE | 0 | 0 | 1
  Any SAE leading to study discontinuation | 0 | 0 | 0
  Any SAE related to the study treatment | 0 | 0 | 0
  Any SAE related to the challenge virus | 0 | 0 | 1
  Any death | 0 | 0 | 0

22. Secondary Outcome: Immunogenicity: Number of Participants Positive for Anti-palivizumab Antibody (ADA)
Description: Determination of the incidence of anti-palivizumab ADA (number and percent of participants tested positive for anti-palivizumab ADA). ADA positive participant: baseline negative and any sample after treatment positive, or baseline positive and titre increased 4- to 9-fold after treatment) before the dose of palivizumab and at scheduled post-dose assessments.
Time Frame: Part 2: prior to infusion with Palivizumab and 7, 13, and 29 days post Palivizumab infusion.
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Palivizumab (Synagis™) (Part 2)
Number analyzed (Participants) | 25
Participants | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 28
Description: Adverse events were coded using the most current version of the Medical Dictionary for Regulatory Activities (MedDRA) and summarized by system organ class, preferred term, and treatment group for the number of AEs reported and the number and percentage of patients reporting each AE.
Arm/Group | Double-blind Placebo (Part 2) | Double-blind Palivizumab (Synagis™) (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 12/25 | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Placebo (Part 2) (N=25) | Double-blind Palivizumab (Synagis™) (Part 2) (N=25)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) — Considered by the investigator to be probably related to challenge virus inoculation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Placebo (Part 2) (N=25) | Double-blind Palivizumab (Synagis™) (Part 2) (N=25)
Alanine Aminotransferase Increased (Investigations) | 6 (6) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is >60 days but < or= 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication if it does not include any reference to the Sponsor, any Study Identifier, or any Property or other Confidential Information of the Sponsor, other than the anonymized Non-drug data.

DOCUMENTS (2):
  • Study Protocol (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT04540627/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT04540627/SAP_001.pdf